CLINICAL TRIAL: NCT05797961
Title: HIV Self-testing With Online Supervision for Vietnamese MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Puerto Rico (Other); US Military HIV Research Program (Network); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH123337 (NIH); R34MH123337 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to either HIV testing with online supervision or venue testing as usual
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV self-testing with online supervision (Experimental): HIV self-testing with online supervision
  Interventions: Behavioral: HIV self-testing with online supervision
- Control (Other): venue-based HIV testing
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: HIV self-testing with online supervision — A pilot study to assess the feasibility of HIV self-testing with online supervision
  Arms: HIV self-testing with online supervision
Other: Control — venue-based HIV testing
  Arms: Control

SUMMARY:
Although global rates of HIV infection have decreased overall, rates among men who have sex with men (MSM) in Southeast Asia are increasing. A recent review of available global data and the molecular epidemiology of HIV among MSM in Southeast Asia suggests that targeted interventions for MSM populations are necessary to reduce HIV incidence in the region. For example, in Vietnam's urban centers, the HIV epidemic among MSM is growing rapidly, with an estimated prevalence of 17% in Ho Chi Minh City and an estimated incidence of 5.8% among young men who have sex with men in Hanoi. Behavioral epidemiology has also been well-described, with high rates of unprotected sex, multiple concurrent partners, untreated STIs, and poor engagement in the HIV care continuum, including low rates of HIV testing, all contributing to high levels of circulating virus among MSM risk networks.

DETAILED DESCRIPTION:
HIV rates among MSM in Vietnam have increased sharply since 2006. By 2011, rates had reached 19%, with HCMC accounting for the largest number of infections. MSM, particularly YMSM, continue to have low rates of HIV testing and poor engagement in HIV care. Studies have identified various risk factors, including low knowledge and perceived risk, sexual risk and STIs/HIV, complexity in identity and meaning, substance use and mental health, limited HIV interventions, and poor engagement in health services. Increasing HIV testing among MSM, particularly YMSM, is crucial for early detection and enrolment in ART. However, individual and institutional-level barriers hinder testing, such as poor knowledge, stigma, and poor repeat testing. Using the internet as an intervention platform can reach and engage MSM who cannot be reached using conventional health-engagement approaches.

The proposed study aims to adapt and pilot test an online HIV testing intervention (OHT) targeted at young men who have sex with men (MSM) in Ho Chi Minh City, Vietnam. The OHT intervention was developed and successfully implemented among MSM in Thailand, showing significant impacts on testing rates and linkage to HIV care. The proposed study builds on longstanding collaborations between HIV researchers from Mahidol University in Thailand and a local community-based organization that serves YMSM in Vietnam. The findings from the proposed study will have important implications for assessing the potential for OHT intervention to overcome profound and longstanding barriers to HIV testing among YMSM in Vietnam, an outcome that if brought to scale could significantly improve enrolment in ART and reduce HIV incidence. Innovative strategies to increase testing and improve continuum will be needed to reduce HIV transmission in Vietnam, where little data is available on uptake of HIV testing among Vietnamese MSM, and a high proportion of men who have sex with men surveyed have never been voluntarily tested for HIV. HIV self-testing with online supervision represents an important strategy to improve scale-up of HIV testing among Vietnamese MSM. The proposed OHT can overcome the barrier of face-to-face testing and counseling, while ensuring that Vietnamese YMSM receive real-time guidance and support for self-testing and linkage to care and treatment, if positive.

The project's aims are: (1) to conduct a qualitative study with Focus Group Discussions (FGDs) to identify potential barriers and facilitators to the uptake of OHT among YMSM in HCMC; (2) to conduct a quantitative study with online survey questionnaires to adapt the existing Thai OHT intervention for use among YMSM in Vietnam, including translation and socio-cultural refinement of testing kits, clip video content, online pre-and post-test counseling, and broader socio-cultural contexts. Data from Aim 1 will be analyzed and used to design the test kit, the clip video content, and when and how the HIV counselor will conduct pre-and post-test counseling. Moreover, willingness to engage in OHT as well as factors related to sustained testing will be collected through an online survey, and (3) to conduct a pilot study with Randomized Control Trial to demonstrate the feasibility and acceptability of the adapted OHT intervention, including the use of an HIV rapid diagnostic antibody/antigen-based self-testing with an HIV counselor through video conferencing. YMSM recruited through the online survey who indicated an interest in OHT will be randomly selected to the OHT group or the venue-based testing group (standard of care), using repeated measures at 6 and 12 months to compare HIV testing rates and behavioral outcomes because of retention and we need to understand how the socio-cultural factors affecting to OHT retention.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-29 years at cohort baseline
* Self-reported male gender
* Self-reported having had anal sex with another man in the past 12 months
* Speak, read and write Vietnamese
* Vietnamese citizenship
* Resident of the assessment city (Ho Chi Minh City) for at least 6 months

Exclusion Criteria:

* Do not consent to HIV self-testing with online supervision
* Not willing to give contact information for follow-up assessments

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Guadamuz, PhD, Principal Investigator — Mahidol University; Giang M Le, MD, Study Chair — Hanoi Medical University
Locations (1):
- Center for Applied Research on Men and Health (CARMAH), Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited over one year using online and offline outreach to reach YMSM in Ho Chi Minh City. Online recruitment will use social media, NGO networks, and youth networks. All survey respondents will receive a mobile top-up worth approximately 2 USD. Interested individuals will complete online eligibility screening and provide electronic informed consent (e-consent). Those testing HIV-positive will not join the pilot. The pilot will recruit 100 YMSM, randomized into a 50-person
Groups:
- HIV Self-testing With Online Supervision: Participants receive an HIV self-testing kit delivered to their home and complete the test with real-time online counselling and supervision by a nurse via Zalo. The nurse provides pre-test counselling, guides proper use of the kit, assists with result interpretation, and ensures confidentiality throughout the process.
Period: Overall Study
Arm/Group | HIV Self-testing With Online Supervision | Control
Started | 50 | 50
Completed 6 Months Follow-up | 46 | 48
Completed 12 Months Follow-up | 45 | 49
Completed | 45 | 49
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Self-testing With Online Supervision | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (3.4) | 24.3 (3.2) | 24.2 (3.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males who have sex with Men | 47 | 47 | 94
  Bisexual Males | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Vietnamese | 50 | 50 | 100
Region of Enrollment [Number; unit: Participants]
  Vietnam | 50 | 50 | 100
Self-Reporteed Last HIV Testing Data [Count of Participants; unit: Participants]
  Never tested | 2 | 2 | 4
  More than 12 months ago | 9 | 3 | 12
  7-12 months ago | 6 | 1 | 7
  ≤ 6 months ago | 33 | 44 | 77
Condom use at last anal intercourse [Count of Participants; unit: Participants] — Used condoms for the entire duration
  Participants | 28 | 21 | 49
Participation in group sex activities (ever) [Count of Participants; unit: Participants] | 19 | 17 | 36
Participant has given or received items or opportunities in exchange for sex [Count of Participants; unit: Participants]
  Yes, I was the one receiving money, things, opportunities and so on | 2 | 4 | 6
  Yes, I was the one giving money, things, opportunities and so on | 2 | 0 | 2
  Yes, I have both given and received money, things, opportunities and so on | 2 | 6 | 8
  No | 44 | 40 | 84
Depression (CES-D-10) [Count of Participants; unit: Participants] — Measure Description: Depression was assessed using the 10-item Center for Epidemiologic Studies Depression Scale (CES-D-10), a validated screening tool for depressive symptoms. Each item is rated on a 4-point Likert scale ranging from 0 ("Rarely or none of the time") to 3 ("All of the time"). The total score ranges from 0 to 30, with higher scores indicating more severe depressive symptoms. A total score of ≥10 was used as the cut-off to classify participants as having depression. The reported outcome reflects the number and percentage of participants meeting this cut-off.
  Participants | 27 | 27 | 54
Risk of Suicide (SBQ-R) [Count of Participants; unit: Participants] — [1]Measure Description: Suicidal risk was assessed using the Suicide Behaviors Questionnaire-Revised (SBQ-R), a validated screening tool for suicidal thoughts and behaviors. The SBQ-R includes 4 items assessing (1) lifetime suicidal ideation and/or attempts, (2) frequency of suicidal ideation in the past 12 months, (3) threats of suicide attempts, and (4) self-reported likelihood of future suicidal behavior. Total scores range from 3 to 18, with higher scores indicating greater risk. Participants with a total score of ≥7 were classified as being at risk of suicide. The reported outcome reflect
  Participants | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: HIV Self-testing With Online Supervision Past 6 Months at Baseline
Description: Number of participants who have gone through the intervention (self-tested for HIV with online supervision past 6 months). For the control group, participants will answer a yes/no question if they have tested for HIV in the past 6 months.
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 50 | 50
Participants | 50 | 44

2. Secondary Outcome: Prevalence of HIV Positive Among YMSM at Baseline
Description: Number of participants who are HIV-positive. For the intervention group (participants who performed HIV self-testing with online supervision in the past 6 months), HIV status is obtained from the supervised self-test results. For the control group, participants report their HIV status through the survey, based on whether they had an HIV test in the past 6 months.
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 50 | 50
Participants | 2 | 0

3. Secondary Outcome: Prevalence of HIV Positive Among YMSM at 6 Months
Description: as for outcome 2
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 46 | 48
Participants | 0 | 1

4. Primary Outcome: HIV Self-testing With Online Supervision Past 6 Months at 6 Months
Description: as for outcome 1
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 46 | 48
Participants | 46 | 38

5. Primary Outcome: HIV Self-testing With Online Supervision Past 6 Months at 12 Months
Description: as for outcome 1
Time Frame: Assessed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 45 | 49
Participants | 45 | 35

6. Secondary Outcome: Prevalence of HIV Positive Among YMSM at 12 Months
Description: as for outcome 2
Time Frame: Assessed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 45 | 49
Participants | 0 | 2

7. Secondary Outcome: HIV Incidence/Seroconversion at Baseline
Description: Number of participants with new HIV infections (seroconversion) during each follow-up period, reported as the number of cases. HIV status in the intervention group is obtained from supervised HIV self-testing, while in the control group it is self-reported through the survey.
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 50 | 50
Participants | 2 | 0

8. Secondary Outcome: HIV Incidence/Seroconversion at 6 Months
Description: as for outcome 7
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 46 | 48
Participants | 0 | 1

9. Secondary Outcome: HIV Incidence/Seroconversion at 12 Months
Description: as for outcome 7
Time Frame: Assessed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-testing With Online Supervision | Control
Number analyzed (Participants) | 45 | 49
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From baseline to 12 months
Arm/Group | HIV Self-testing With Online Supervision | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT05797961/Prot_SAP_ICF_000.pdf